CLINICAL TRIAL: NCT04461119
Title: A Phase II, Randomized, 4-Week, Double-Blind, Placebo-Controlled, Multiple-Dose Study, Designed to Determine the Safety, Tolerability, EEG Effects and Preliminary Efficacy of Fixed Oral Doses of 7.5 and 15 MG BID of Evenamide in Patients With Chronic Schizophrenia Who Are Symptomatic on Their Current Second-Generation Antipsychotic Medication
Brief Title: Study to Determine the Safety, Tolerability, and Efficacy of Evenamide in Patients With Chronic Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-3509/008/II/2019
Record Dates: First submitted 2020-06-19; First posted 2020-07-08 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Evenamide 7.5 mg bid (Experimental): Evenamide capsules 7.5 mg BID for a total of 28 dosing days
  Interventions: Drug: Evenamide
- Evenamide 15 mg bid (Experimental): Evenamide capsules 15.0 mg BID for a total of 28 dosing days
  Interventions: Drug: Evenamide
- Placebo (Placebo Comparator): Matching placebo capsules BID for a total of 28 dosing days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evenamide — oral capsules for 4 weeks of treatment
  Other Names: NW-3509
  Arms: Evenamide 15 mg bid; Evenamide 7.5 mg bid
Drug: Placebo — oral capsules for 4 weeks of treatment
  Arms: Placebo

SUMMARY:
This 4-week study will evaluate the safety, tolerability and preliminary evidence of efficacy of evenamide (7.5,and 15 mg and placebo, bid) treatment in outpatients with chronic schizophrenia.

DETAILED DESCRIPTION:
This is a prospective, 4-week, randomized, double-blind, placebo-controlled, study designed to evaluate the safety, tolerability, EEG effects, and preliminary efficacy of two fixed oral doses of evenamide of 7.5 mg and 15 mg bid (15 and 30 mg/day) in outpatients with chronic schizophrenia who are receiving treatment at constant doses of one of the following atypical antipsychotics: aripiprazole, clozapine, quetiapine, olanzapine, paliperidone or risperidone. Approximately 120 patients will be randomized in a 1:1:1 ratio to receive either evenamide 7.5 or 15 mg, or placebo, given bid.

ELIGIBILITY:
Inclusion Criteria:

Demographics

* Age - 18 years, or older
* Sex - male, or non-childbearing potential female unless practicing adequate contraception

Psychiatric

* Has a current diagnosis of schizophrenia in accordance with DSM-5.
* Has been treated with antipsychotics for at least 2 years.
* Has a total score on the PANSS < 80.
* Has a Clinical Global Impression - Severity of disease (CGI-S) rating of mildly, moderately or moderately severely ill (score of 3, 4 or 5).
* Needs antipsychotic treatment and is currently receiving a stable dose (minimally for 4 weeks prior to screening) of aripiprazole, clozapine, quetiapine, olanzapine, paliperidone, or risperidone (at least 2 mg risperidone dose-equivalent)
* Current symptoms have been stably present for at least one month

Procedural

* Patient resides at home or in a residential care facility
* If taking clozapine, patient agrees to blood monitoring

Exclusion Criteria:

Psychiatric

* Severity of current episode of psychosis requires that the patient be hospitalized. Patients who are chronically hospitalized or in psychiatric day-care, whose hospitalization is for logistic reasons and not due to the severity of their illness, will be eligible for the study.
* Severity of psychosis is rated severe or higher (CGI-S of 6 or greater).
* Known suicidal risk. A "yes" response on the C-SSRS Suicidal Ideation Item 4 or Item 5, or a "yes" response on any of the five C-SSRS Suicidal Behavior items, at screening, or a suicide attempt within the past 6 months, excludes the patient from the study.
* Patients with a diagnosis of Treatment resistance
* History of neuroleptic malignant syndrome, priapism.
* Current moderate or severe tardive dyskinesia.

Medical Status

* Abnormal epileptiform phenomena (3 per second spike and slow wave discharges) observed on screening EEG. History or current diagnosis of epilepsy or seizure disorder (other than febrile seizures in childhood)
* Insulin-dependent diabetes mellitus
* History or current diagnosis of any neurodegenerative illnesses
* Loss of 500 ml or more of blood during the 3-month period before study enrollment, e.g. as a donor

Cardiovascular

* A current diagnosis of severe or unstable cardiovascular disease
* Any clinically significant ECG abnormality
* Abnormal vital signs

Laboratory abnormalities

* Clinically significant abnormalities in routine laboratory examinations
* History and/or presence of hepatitis B and/or C
* Positive results from the HIV serology.
* Positive results of the drug and alcohol tests
* Clinically significant or unstable hypothyroidism or hyperthyroidism

Concomitant therapy

* Treatment with SSRIs that are moderate/potent inhibitors of CYP2D6 (e.g. fluoxetine)
* Treatment with drugs capable of inducing/inhibiting hepatic enzyme metabolism
* Current treatment with sodium channel blockers
* Exposure to any investigational drug within 5 weeks or 5 half-lives (whichever is longer) prior to screening
* A known exaggerated pharmacological sensitivity or hypersensitivity to drugs similar to evenamide (e.g. lamotrigine, carbamazepine, oxcarbazepine, topiramate, etc.), or any components of the evenamide or matching placebo capsules
* Treatment with a drug or treatment known to cause major organ system toxicity, e.g. tamoxifen, within 4 weeks, or received radiation therapy or a drug with cytotoxic potential, e.g. chemotherapy, during the past year
* Electroconvulsive therapy (ECT) or treatment with a transcranial magnetic stimulation (TMS) device within 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability - incidence of Treatment-Emergent Adverse Events [TEAEs], Serious Adverse Events [AEs], and Adverse Events leading to discontinuation [ADOs] | 4 Week study
  Comparison will be made between the evenamide and placebo groups in the proportion of patients experiencing Serious Adverse Events [SAEs], Adverse Events leading to discontinuation [ADOs] and, Treatment-Emergent Adverse Events [TEAEs].
Change from baseline in Positive and Negative Syndrome Scale [PANSS] total score | 4 Week study
  Efficacy measure of mean change from baseline to endpoint of Positive and Negative Syndrome Scale [PANSS] total score: this is a 30-item scale that was designed to assess various symptoms of schizophrenia each rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology).

SECONDARY OUTCOMES:
Key secondary - Change from baseline in clinical global impression severity of Illness [CGI-S] score | 4 Week study
  Efficacy measure by mean change from baseline top endpoint of the Clinical Global Impression Severity of Illness [CGI-S]: the investigator rates the severity of a subject's condition on a 7-point scale ranging from 1 (no symptoms) to 7 (very severe).
Rating at endpoint on the CGI - Change from baseline (CGI-C) | 4 Week study
  Efficacy measured by Clinical Global Impression of Change [CGI-C]: 7-point scale requiring the clinician to rate how much the patient's illness has improved at endpoint relative to the baseline state (score of 1, 2, 3); CGI-C ranges from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating "no change".
Evaluate plasma drug concentrations over time for evenamide and its major metabolite, (3-butoxy-phenyl)-acetic acid | 4 Week study
  Determine the multiple-dose plasma concentrations of evenamide and its major metabolite, (3-butoxy-phenyl)-acetic acid, at the doses tested.
  Doses of evenamide to be evaluated in this study, compared to placebo, will be 7.5 mg bid, and 15 mg bid, with key information being collected at or near the time of the predicted maximal plasma concentration (Tmax) for evenamide.
Comparison of plasma drug concentrations over time for evenamide and its major metabolite, (3-butoxy-phenyl)-acetic acid between the dosing arms 7.5 mg BID and 15.0 mg BID | 4 Week study
  Determine if the PK parameters are dose proportional. Doses of evenamide to be evaluated in this study, compared to placebo, will be 7.5 mg bid, and 15 mg bid, with key information being collected at or near the time of the predicted maximal plasma concentration (Tmax) for evenamide.
Efficacy - changes in daily functioning | 4 Week study
  Determine the effect of evenamide, compared to placebo, on daily functioning, based on changes on the Strauss-Carpenter Level of Functioning (LOF) scale; The LOF is a semi-structured, clinician-administered scale of nine items. The individual items fall into four domains, with higher scores on a 5-point scale (0 - 4) reflecting better functioning. The subscales are Social Contacts (frequency and quality of social contacts), Work (quantity and quality of useful work), Symptomatology (absence of symptoms and recent hospitalization), and Function (ability to meet basic needs, fullness of life, and overall level of function). A total score is calculated as the sum of the raw scores across the nine items.
Efficacy - rating score of patient satisfaction with the study medication | 4 Week study
  Determine the patient's satisfaction with the study medication, compared to their previous treatment, based on improvements on the Medication Satisfaction Questionnaire (MSQ) which is a single-item, 7-point Likert-type scale for patients with schizophrenia to rate their satisfaction with their antipsychotic medication.
  The patient's response to the question "Overall, how satisfied are you with your current antipsychotic medication(s)?" is rated by the clinician as follows: 1 = extremely dissatisfied, 2 = very dissatisfied, 3 = somewhat dissatisfied, 4 = neither satisfied nor dissatisfied, 5 = somewhat satisfied, 6 = very satisfied, and 7 = extremely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Anand, MD, Study Director — Newron Pharmaceuticals
Locations (14):
- United States (3):
  - Behavioral Research Specialists, LLC, Glendale, California
  - CBH Health, LLC, Gaithersburg, Maryland
  - Community Clinical Research CCR, Austin, Texas
- India (11):
  - Help Hospitals Clinical Research Department, Vijayawada, Andhra Pradesh
  - St. John's Medical College Hospital, Koramangala, Karnataka
  - Mangala Hospital and Mangala Kidney Foundation, Department of Psychiatry, Mangalore, Karnataka
  - IQRAA Psychiatry Care and Rehabilitation Centre, Kozhikode, Kerala
  - Deenanath Mangeshkar Hospital Research Center, Pune, Maharashtra
  - Sujata Birla Hospital, Pune, Maharashtra
  - Post Graduate Institute of Medical Education and Research, Chandigarh, Punjab
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Sri Ramachandra Medical College, Department of Psychiatry, Chennai, Tamil Nadu
  - Ahana Hospital LLP, Madurai, Tamil Nadu
  - Asha Hospital, Hyderabad, Telangana